CLINICAL TRIAL: NCT01537536
Title: An Open-label Phase II Trial Evaluating the Efficacy and Safety of Neoadjuvant EndoTAG-1 in Combination With Paclitaxel in Patients With HER2-negative Breast Cancer
Brief Title: Trial of Neoadjuvant EndoTAG-1 in Combination With Paclitaxel in HER2-negative Breast Cancer
Acronym: EndoTAG-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IJBNeoEndoTAG-1
Record Dates: First submitted 2011-09-20; First posted 2012-02-23 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2012-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Neoadjuvant chemotherapy; EndoTAG-1
MeSH Terms: conditions — Breast Neoplasms | interventions — MBT-0206

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EndoTAG-1 (Experimental): Weekly treatment with EndoTAG-1 (22 mg/m2) plus paclitaxel (70 mg/m2) for 12 weeks (ET+P) followed by subsequent treatment with the standard FEC regimen (Fluorouracil 500 mg/m2, Epirubicin 100 mg/m2, Cyclophosphamide 500 mg/m2) once every 3 weeks for 3 cycles of therapy followed by surgery.
  Interventions: Drug: EndoTAG-1

INTERVENTIONS:
Drug: EndoTAG-1 — EndoTAG-1 (22 mg/m2 liposomal paclitaxel) + Paclitaxel (70 mg/m2) Weekly i.v. infusions of EndoTAG-1 and paclitaxel for 12 weeks followed by subsequent treatment with the standard FEC regimen (Fluorouracil 500 mg/m2, Epirubicin 100 mg/m2, Cyclophosphamide 500 mg/m2) once every 3 weeks for 3 cycles of therapy followed by surgery.
  Other Names: Non applicable

SUMMARY:
The study hypothesis is that the new drug EndoTAG-1 will improve tumor volume reduction as measured by Magnetic Resonance Imaging when added to a standard chemotherapy regimen of weekly paclitaxel. This is a prospective single-center study that will investigate the activity of EndoTAG-1 + paclitaxel combination therapy in patients with HER2-negative breast cancer that are candidate for receiving chemotherapy before surgery (neoadjuvant chemotherapy).

DETAILED DESCRIPTION:
This is a prospective, single-center, open-label phase II clinical trial investigating the activity of EndoTAG-1 + paclitaxel combination therapy in patients with HER2-negative BC candidate for neoadjuvant chemotherapy, as measured by the decrease in MRI-estimated tumour volume at the end of EndoTAG-1 + paclitaxel administration. Patients will be stratified by hormone receptor status.

A total of 20 female patients with non-metastatic HER2-negative breast cancer candidate for neoadjuvant chemotherapy and meeting all study eligibility criteria will receive 12 weekly infusions of EndoTAG-1 (22 mg/m2 liposomal paclitaxel) in combination with paclitaxel (70 mg/m2) followed by 3 cycles of FEC (Fluorouracil 500mg/m2, Epirubicin 100mg/m2, Cyclophosphamide 500mg/m2) every 3 weeks (experimental group) The study hypothesis is that EndoTAG-1 will improve MRI- estimated volume reduction when added to weekly paclitaxel. The null hypothesis is that combination has no or a negligible effect on volume reduction (defined as lower or equal to a 50% decrease) versus the alternative hypothesis that the combination yields at least a 80% average decrease in MRI- estimated volume at the end of weekly paclitaxel and EndoTAG-1 administration from baseline

ELIGIBILITY:
Inclusion Criteria:

1. newly diagnosed histologically confirmed BC with breast infiltrating carcinoma of histological grade > 1 (either operable, or locally advanced or inflammatory) candidate for neoadjuvant chemotherapy
2. HER2-negative tumor, defined according to immunohistochemistry or using fluorescent in-situ hybridization (FISH)
3. ECOG performance status 0 or 1
4. Gender: female
5. Age : >= 18 years old
6. Negative pregnancy test (females of childbearing potential)
7. Willingness to perform double-barrier-contraception during study and for 6 months post chemotherapy treatment (females of childbearing potential)
8. Signed informed consent

Exclusion Criteria:

1. Metastatic or relapsed disease
2. Major surgery < 3 weeks prior to enrollment
3. Severe pulmonary obstructive or restrictive disease
4. Uncontrolled inflammatory disease (autoimmune or infectious)
5. Clinically significant cardiac disease (NYHA stadium > 2)
6. Results of laboratory tests (hematology, chemistry) outside specified limits:

   * WBC ≤ 3 x 109/L
   * ANC < 1.5 x 109/L
   * Platelets < 100 x 109/L
   * Hb ≤ 9.0 g/dl (≤ 5.6 mmol/l)
   * PTT/ INR > 1.5 x ULN
   * AST or ALT > 2.5 x ULN
   * Alkaline Phosphatase > 2 x ULN
   * Total Bilirubin > 1.5 x ULN
7. Pregnancy or nursing status
8. Known positive HIV testing
9. Known hypersensitivity to any component of the EndoTAG-1, paclitaxel or FEC formulations
10. History of malignancy other than breast cancer < 5 years prior to enrollment, except skin cancer (i.e. basal or squamous cell carcinoma) treated locally
11. History of active or significant neurological disorder or psychiatric disorder that would prohibit the understanding and giving of informed consent, or would interfere in the clinical and radiological evaluation of central nervous system during the trial
12. Concurrent treatment with other experimental products. Participation in another clinical trial with any investigational product within 30 days prior to study entry

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
MRI-estimated tumour volume at the end of neoadjuvant EndoTAG-1 + paclitaxel administration vs. baseline. | 15 weeks after start of neoadjuvant chemotherapy.
  To investigate the activity of EndoTAG-1 + paclitaxel combination therapy in patients with HER2-negative BC candidate for neoadjuvant chemotherapy, as measured by the decrease in MRI-estimated tumour volume at the end of neoadjuvant EndoTAG-1 + paclitaxel administration vs. baseline.

SECONDARY OUTCOMES:
Rate of pathological complete response (pCR). | 27 weeks after start of neoadjuvant chemotherapy.
  Rate of pathological complete response (pCR) at the end of neo-adjuvant chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Michail Ignatiadis, MD, PhD, Principal Investigator — Jules Bordet Institute
Locations (1):
- Institut Jules Bordet, Brussels, Brussels Capital, Belgium

REFERENCES:
- [Derived] Ignatiadis M, Zardavas D, Lemort M, Wilke C, Vanderbeeken MC, D'Hondt V, De Azambuja E, Gombos A, Lebrun F, Dal Lago L, Bustin F, Maetens M, Ameye L, Veys I, Michiels S, Paesmans M, Larsimont D, Sotiriou C, Nogaret JM, Piccart M, Awada A. Feasibility Study of EndoTAG-1, a Tumor Endothelial Targeting Agent, in Combination with Paclitaxel followed by FEC as Induction Therapy in HER2-Negative Breast Cancer. PLoS One. 2016 Jul 25;11(7):e0154009. doi: 10.1371/journal.pone.0154009. eCollection 2016. PMID 27454930